CLINICAL TRIAL: NCT06814756
Title: Bacteriophage Therapy for Morganella Morganii Prosthetic Joint Infection
Acronym: PHAGE-MOM-001
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Qeen Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB25-0157
Record Dates: First submitted 2025-01-22; First posted 2025-02-07 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-01

CONDITIONS: Prosthetic Joint Infections of Hip
Keywords: Bacteriophage; Periprosthetic joint infection; Phage therapy
MeSH Terms: interventions — Phage Therapy

STUDY DESIGN:
Intervention Model Description: Single patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label Arm (Experimental): Bacteriophage drug product
  Interventions: Biological: phage therapy

INTERVENTIONS:
Biological: phage therapy — Single anti-Morganella morganii bacteriophage drug product

SUMMARY:
This is a single-patient, phase I/II clinical trial that aims to evaluate the potential of a bacteriophage drug product to treat and prevent the recurrence of a Morganella morganii prosthetic joint infection of the hip. The patient has exhausted all conventional therapies, both surgical and medical, at considerable detriment to their quality of life. The treatment involves 2 intra-articular injections of bacteriophages into the joint and surrounding area and 14 days of intravenous phage therapy. The goal is to eliminate the infection and prevent further complications, providing a potential new treatment avenue for patients with difficult-to-treat infections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active chronic prosthetic joint infection
* Causative bacteria is susceptible to bacteriophage therapy in vitro
* History of multiple failed antibiotic and surgical interventions

Exclusion Criteria:

* Stage 5 chronic kidney disease
* Cirrhosis
* A known allergy to phage products
* Fever
* Involvement in another clinical trial
* Pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Clinical response to phage therapy as determined by participant's absence of physical symptoms | 1 year
  Resolution of the infection, indicated by the absence of clinical symptoms such as wound drainage, swelling, erythema, pain, and fever. This will be determined by a questionnaire and monthly assessments by a Infectious Disease physician.

SECONDARY OUTCOMES:
Safety and tolerability of phage therapy determined by incidence of treatment-emergent adverse events | 29 days
  The safety outcome focuses on monitoring and documenting any adverse events (both serious and not) or reactions associated with bacteriophage therapy. Key safety measures include observing for immediate allergic reactions during the first dose, conducting regular clinical assessments, and performing routine bloodwork to detect any potential organ damage or unexpected side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Centre, University of Calgary, Calgary, Canada

IPD SHARING:
Plan to Share IPD: No